CLINICAL TRIAL: NCT02701842
Title: ImPACT Online Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImPACT Applications, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: QPR-16-05
Record Dates: First submitted 2016-02-27; First posted 2016-03-08 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Brain Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Validity (Experimental): ImPACT Online a computerized test will be administered to subjects. They will also receive a battery of paper and pencil neuropsychological tests.
  Interventions: Device: ImPACT Online/Paper Pencil Tests
- Test/Re-Test (Active Comparator): ImPACT Online will be administered at 2 time points.
  Interventions: Device: ImPACT Online

INTERVENTIONS:
Device: ImPACT Online/Paper Pencil Tests
  Arms: Validity
Device: ImPACT Online
  Arms: Test/Re-Test

SUMMARY:
The researchers want to find out more about a standalone software application, ImPACT Online and how it relates to other commonly used tests of memory, attention and reaction time. ImPACT Online is a computer-based neurocognitive test for concussion management. The test was designed to help measure the effects of concussion on cognitive processes (for example, memory, attention, brain speed) and visual functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-59
* Primary English speaking or fluent in English.
* No known special education diagnosis excluding a 504 designation.
* Currently not suffering from a concussion or being treated for a concussion.
* No known physical or psychological impairment that would affect their ability to perform the test.
* An average or above average score on the RIST (Reynolds Intellectual Screening Test).

Exclusion Criteria:

* Documentation of a known special education diagnosis other than a 504 designation.
* English is not their primary language nor are they proficient in the English language.
* Currently suffering from a concussion or being treated for a concussion.
* A below average score on the RIST.

Ages: 12 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Validity is established through correlation studies with well-known measures of memory and processing speed. | 12 Months
Reliability will be established through a test/re-test to establish results should be stable over time. | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- ImPACT Applications Inc., Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No